CLINICAL TRIAL: NCT01417403
Title: A Phase 1 Study of Hydroxychloroquine in Patients With Solid Tumors Receiving Radiotherapy for Bone Metastases
Brief Title: Hydroxychloroquine in Treating Patients With Solid Tumors Undergoing Radiation Therapy for Bone Metastases
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Recently published data that has shown HCQ to be safe when combined with chemo and or radiation at even higher doses than what is used in this study.
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-13713; NCI-2011-02310 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA016059 (NIH)
Record Dates: First submitted 2011-08-10; First posted 2011-08-16 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Bone Metastases; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Hydroxychloroquine; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (radiosensitization therapy) (Experimental): Beginning 3 days before the initiation of radiotherapy, patients receive hydroxychloroquine PO QD or BID. Treatment continues until completion of radiotherapy.
  Interventions: Drug: hydroxychloroquine; Radiation: radiation therapy

INTERVENTIONS:
Drug: hydroxychloroquine — Given PO
  Other Names: HCQ
Radiation: radiation therapy — Undergo radiotherapy
  Other Names: irradiation; radiotherapy; therapy, radiation

SUMMARY:
This phase I trial studies the side effects and best dose of hydroxychloroquine in treating patients with solid tumors undergoing radiation therapy for bone metastases. Drugs, such as hydroxychloroquine, may make tumor cells more sensitive to radiation therapy

DETAILED DESCRIPTION:
OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of hydroxychloroquine that can safely be administered to cancer patients in association with radiation prior to developing this approach for disease treatment.

OUTLINE: This is a dose escalation study.

Beginning 3 days before the initiation of radiotherapy, patients receive hydroxychloroquine orally (PO) once daily (QD) or twice daily (BID). Treatment continues until completion of radiotherapy.

After completion of study treatment, patients are followed up at 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed solid tumor with radiographic evidence of bony metastatic disease and symptoms requiring palliative radiotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 6 weeks
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin =< 1.5 X institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =<2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with calculated creatinine levels above institutional normal limits
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy within 4 weeks prior to entering the study or those who have not recovered from acute adverse events due to agents administered more than 4 weeks earlier
* Patients may not have received prior radiotherapy to the intended site
* Patients who have not recovered from acute adverse events due to previous radiotherapy
* Patients may not be receiving any other investigational agents
* Patients who are neurologically unstable due to uncontrolled brain metastases are excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. - - History of allergic reactions attributed to compounds of similar chemical or biologic composition to hydroxychloroquine
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients who are pregnant or may become pregnant during treatment
* Patients with severe psoriasis who may experience a flare of disease with hydroxychloroquine use
* Patients with known liver dysfunction (elevated transaminases or abnormal coagulation studies); patients with metastatic disease to the liver with normal liver function studies may be enrolled
* Patients with retinopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
MTD of hydroxychloroquine that can be safely administered to cancer patients in association with radiotherapy | 12 weeks
  Safety assessments weekly during treatment and at 4 weeks post-radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Cuttino, Principal Investigator — Massey Cancer Center
Locations (1):
- Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia, United States

REFERENCES:
- See also: VCU Massey Cancer Center — http://www.massey.vcu.edu/